CLINICAL TRIAL: NCT05950620
Title: Pilot and Feasibility Project to Establish a Childhood Nutrition and Health Clinic Managing Weight and Obesity Complications in a Primary Care Pediatric Practice
Brief Title: Bringing Weight Management Into the Primary Care Pediatric Practice
Status: Recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: William H. Hurt Foundation (Unknown)
Responsible Party: Principal Investigator, Jonathan Purnell, Professor, Oregon Health and Science University
Other Study IDs: IRB 24927
Record Dates: First submitted 2023-07-11; First posted 2023-07-18 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention: Pediatric patients with obesity or in need of weight management for unwanted weight gain.
  Interventions: Other: Medical obesity management.
- Controls: Historic controls matched to the Intervention group on age, sex, and BMI percentile.

INTERVENTIONS:
Other: Medical obesity management. — Dietician visits, education, anti-obesity medications, and/or referral for metabolic-bariatric surgery as indicated by American Academy of Pediatrics guidelines for obesity management.
  Groups: Intervention

SUMMARY:
This project aims to move what is currently a specialty-care model for the management of obesity of children and adolescents into the primary care setting.

DETAILED DESCRIPTION:
The goal of this project is to create a sustainable clinical model in the primary care setting that improves nutritional health, lessens obesity, and addresses weight-related complications of children and adolescents to reduce risk for metabolic disease in later life. The primary objectives include tracking changes in BMI (both absolute and percentile) and levels of hemoglobin A1c, liver enzymes (AST, ALT levels), and lipids in patients seen in a primary care setting by a general pediatrician board-certified in obesity medicine. Secondary objectives include tracking patient adherence, follow-up, and retention.

ELIGIBILITY:
Inclusion Criteria:

Children with obesity (BMI > 30 kg/m2 or > 95th percentile) or in need of weight management of unwanted weight gain.

Exclusion Criteria:

None.

Ages: 1 Month to 21 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients in a general pediatrician's office internally in Portland, Oregon.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in body weight | Baseline to follow-up (1-3 years)
  Body weight in kg
Change in body height | Baseline to follow-up (1-3 years)
  Body height in meters
Change in BMI | Baseline to follow-up (1-3 years)
  BMI will be calculated using the formula: kg weight / m2 height. Will be in both absolute and percentile for age
Impact on glucose control | Baseline to follow-up (1-3 years)
  Hemoglobin A1c levels
Impact on fatty liver | Baseline to follow-up (1-3 years)
  Levels of liver enzymes ALT, AST
Impact on lipid levels | Baseline to follow-up (1-3 years)
  Levels of total, LDL, HDL, and non-HDL cholesterol. Triglycerides.

SECONDARY OUTCOMES:
Patient follow-up metrics | Baseline to follow-up (1-3 years)
  Patient clinical follow-up rate, medication adherence, and retention

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The Children's Clinic, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No
This study uses anonymized data. No IPD will be generated.